CLINICAL TRIAL: NCT06111001
Title: Single Cohort Pilot Study With NHS Staff to Investigate the Impact on Their Ability to Manage Work Email, Improve Email Productivity, and Digital Wellbeing Before and After Use of the AirEmail v1 Digital Tool in Outlook
Brief Title: NHS Staff Digital Wellbeing Via AirEmail
Acronym: NHS DigiWell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AirEmail Holdings Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022001
Record Dates: First submitted 2023-07-13; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Communication Research; Technostress; Work Related Stress; Burnout, Professional; Well-Being, Psychological
Keywords: Technostress; Technology Related Stress; Healthcare communication; Email communication; National Health Service email; Work Related Stress; Burnout; Well-Being
MeSH Terms: conditions — Occupational Stress; Burnout, Professional; Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Study participants will be enrolled by the NHS Research Coordinator. Participants and their allocation to study groups will not be known to the Sponsor Investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Study Group (Active Comparator): Participants actively using the AirEmail v1 Digital Tool features.
  Interventions: Other: Email use data collection; Other: AirEmail Tips and Tricks training; Other: AirEmail v1 Digital Tool use
- Contemporary Observational Group (Placebo Comparator): Participants whose email use data is collected via the AirEmail v1 Digital Tool
  Interventions: Other: Email use data collection

INTERVENTIONS:
Other: Email use data collection — Participants will initiate the AirEmail v1 Digital Tool. Non-identifiable email use data will be collected.
Other: AirEmail Tips and Tricks training — Participants will watch the "AirEmail Tips and Tricks" training videos ahead of using the AirEmail v1 Digital Tool
  Arms: Active Study Group
Other: AirEmail v1 Digital Tool use — Participants will use the AirEmail v1 Digital Tool features as part of their routine email management in NHSmail, the NHS's Microsoft 365 Outlook platform.
  Arms: Active Study Group

SUMMARY:
The goal of this "digital health intervention" study is to test a novel email management tool called "AirEmail" (version 1, or v1) for its impact on improving key aspects of healthcare email management.

The main questions it aims to answer are:

* What are the effects of technostress in staff employed by the National Health Service (NHS)?
* Can the AirEmail digital tool improve email productivity?
* Can the AirEmail digital tool improve participant digital wellbeing?

Participants will use AirEmail for a period of 4 weeks as part of their routine management of healthcare email. This active use period will be preceded and followed by 2 weeks of an "observational mode" in which email use data is collected.

Researchers will compare participants in the active study group with participants in the contemporary observational group to see if the volume and patterns of email communications have been affected by external factors or AirEmail use.

DETAILED DESCRIPTION:
The NHS DigiWell study is a Before and After Study of a "digital health intervention" testing a novel digital email management tool called "AirEmail" for its impact on improving key aspects of healthcare email management. AirEmail is a Microsoft 365 Outlook registered add-in, a software programme extending the capabilities of, and automating tasks in, Microsoft Outlook.

The study aims to determine the overall effect of the AirEmail Digital Tool over a period of 4 weeks on NHS staff email productivity and digital wellbeing. The active use period will be preceded by 2 weeks of "observational mode" in which email use data will be collected and 2 weeks in which participants will complete induction training. There will be further 2 weeks of "observational mode" following the active period.

Email use statistics data will also be collected from a contemporary observational group for a 10 weeks coinciding with the time period in which active group participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. NHS staff employed at a participating NHS organisation with an active NHS IT account, Microsoft 365 access, and routinely using the Microsoft Outlook app on a computer for email management.
2. Age ≥ 18 years.
3. Able to communicate fluently in English.
4. Have been employed in the same NHS trust for at least 3 months prior to study participation and likely remain employed in the same NHS trust for another at least 3 months.
5. Contracted to work for ≥0.5 full-time equivalent (FTE).
6. Willing to complete study assessments and agree to non-identifiable email usage data being collected for the duration of the study.
7. Currently has (or agrees to create prior to joining the study) ≥500 megabytes of available storage in their NHSmail inbox (the usual total storage capacity of which is 4 gigabytes), and agrees not to exceed their NHSmail storage quota for the duration of the trial to ensure NHSmail performance is not adversely affected by the AirEmail Digital Tool processing and the study data collection.
8. Willing and able to engage IT support to seek resolution of email related issues as required.
9. Meets at least one of the following criteria: a) Receives ≥50 emails a day, or b) sends ≥20 emails a day, or c) spends ≥2 hours in email management on a busy day, in/from their individual inbox, or d) feels dissatisfied with their ability to manage email to an acceptable standard.
10. Willing and able to complete study training activities - estimated to require approximately 45 minutes over a period of maximum 2 weeks - and to configure their email and use the AirEmail v1 features as part of their NHS employment for the duration of the study.

Exclusion Criteria:

1. Currently absent from work for a period lasting, or likely to last, ≥4 weeks, or have returned from long-term absence/leave of ≥4 weeks in ≤4 weeks before joining the study.
2. Plans to take ≥8 working days of Annual Leave coinciding with study participation.
3. Currently participating in another interventional study in the field of digital wellbeing or digital communications.
4. Receives high-volume, high-risk patient-related communication. Note: This would apply for staff employed in clinical pathway coordinator roles, or similar, where even an hour of downtime would compromise patient care.
5. Has any specific accessibility requirements not catered for by the AirEmail v1 application (for example colour blindness which makes seeing highlighted words in Outlook a problem).
6. Relies on using Microsoft Outlook's "categories" feature to manage administrative or clinical workflows.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
Email productivity | 10 weeks
  Self-reported email use productivity
Digital wellbeing | 10 weeks
  Self-reported digital wellbeing

SECONDARY OUTCOMES:
Volume of email activity | 10 weeks
  Number of emails received/sent, their categories and importance
Email use productivity - specific AirEmail features | 10 weeks
  Self reported email use productivity - specific AirEmail features
Digital wellbeing - specific AirEmail features | 10 weeks
  Self-reported digital wellbeing - specific AirEmail features

OTHER OUTCOMES:
Email curation | 10 weeks
  Number/percentage of emails in the curation categories

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mehta, Dr, Principal Investigator — AirEmail Holdings Limited, Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study participants provide consent for sharing anonymized data for the purpose of further research in the field of technostress and digital communications.
Time Frame: Data will be available from 2024
Access Criteria: Any requests related to ethically approved studies in this field will be considered by the Sponsor.

REFERENCES:
- See also: Study website — https://www.nhsdigiwell.com/